CLINICAL TRIAL: NCT01966146
Title: Quantitative Analysis of Catheter-based Interventional Therapies for Treating Valve Insufficiency by Using 3D Echocardiography.
Brief Title: Examination of Valve Insufficiency Before and After MitraClip or TAVI Procedure by 3D Echocardiography Compared to MRI
Acronym: 3D_TTE_TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-067
Record Dates: First submitted 2013-07-17; First posted 2013-10-21 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Development of Standardized Assessment TAVI and MitraClip Procedures by Echocardiography; Aortic Stenosis; Mitral Valve Insufficiency
MeSH Terms: conditions — Aortic Valve Stenosis; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAVI (Experimental): Echocardiography after TAVI
  Interventions: Device: Echography GE Healthcare Vivid E9
- MitraClip (Experimental): Echocardiography after MitraClip procedure
  Interventions: Device: Echography GE Healthcare Vivid E9

INTERVENTIONS:
Device: Echography GE Healthcare Vivid E9 — Echography GE Healthcare Vivid E9

SUMMARY:
Aim of the study is the definition of criteria for a standardized assessment of heart function by 3D echocardiographic procedures. Standardized criteria will be defined to assess aortic valve insufficiency after TAVI and success of mitral valve replacement respectively.

DETAILED DESCRIPTION:
Echocardiography: GE Healthcare Vivid E9

ELIGIBILITY:
Inclusion Criteria:

* patients with severe symptoms of an aortic stenosis who underwent catheter based implantation of an aortic valve
* patients who are planned to undergo a reconstruction of the mitral valve with the MitraClip System
* Patients who are aged above 18 years and legally competent
* signed informed consent

Exclusion Criteria:

* patients with previous myocard infarction, previous heart surgeries, malignity or valvular abnormities > stage 1
* patients with atrial fibrillation
* pregnant and breast-feeding women
* patients with disturbed central nerve system
* patients with pacemaker, implants, ferrous clamps,insulin pump
* patients with tattoo
* patients with claustrophobia
* patiens with asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Quantitative analysis of geometric changes and heart function after heart valve replacement and reconstruction respectively by 3D echocardiographic procedures | Analysis will be performed after heart valve replacement or reconstruction procedures and after 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum RWTH Aachen, Aachen, North Rhine-Westphalia, Germany